CLINICAL TRIAL: NCT03523481
Title: NHF in Acute Hypercapnic Acute Exacerbation of COPD
Status: Completed | Type: Observational
Sponsor: Jens Bräunlich, MD (Other)
Responsible Party: Sponsor-Investigator, Jens Bräunlich, MD, Principal investigator, University of Leipzig
Organization: University of Leipzig (Other)
Other Study IDs: 2
Record Dates: First submitted 2018-04-02; First posted 2018-05-14 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Safety of NHF in Acute Hypercapnic AECOPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NHF use

SUMMARY:
Patients with AECOPD and NIV failure and in absence will be treated with NHF device. Inclusion criteria are pH < 7,38 and pCO2 > 45 mm Hg. Patients were treated if pH >7,38 or refusal of therapy.

ELIGIBILITY:
Inclusion Criteria:

* pH < 7,38
* hypercapnic AECOPD

Exclusion Criteria:

* Need of intubation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AECOPD and failure of NIV therapy
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
pH | up to 24 hours
  Increase in pH

SECONDARY OUTCOMES:
pCO2 | up to 24 hours
  Decrease in pCO2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Germany